CLINICAL TRIAL: NCT02443519
Title: Bronx Mindfulness Based Cognitive Therapy for Migraine: a Randomized Clinical Trial
Brief Title: Bronx MBCT-Migraine
Acronym: BMBCT-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Elizabeth Seng, Assistant Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-4684
Record Dates: First submitted 2015-05-08; First posted 2015-05-14 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Migraine
Keywords: Mindfulness; MBCT; Cognitive Therapy; Disability
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBCT for Migraine (Experimental): In this arm, participants will receive 8 weeks of the manualized treatment Mindfulness Based Cognitive Therapy (MBCT; Day & Thorn). Participants will attend weekly 75-90 minute individual sessions for eight weeks. At each weekly session one of eight broad topics are addressed and discussed (Automatic-Pilot, Dealing with Barriers, Mindfulness of Breath, Staying Present, Allowing/Letting Be, Cognitive Restructuring, Self Care, Application to Headache Pain). Homework is assigned each week, and participants are expected to develop a daily formal mindfulness practice (body scan meditation, seated meditation, breathing meditation, etc). Participants are provided with a course manual, reading materials, and audio recordings to facilitate meditation practice.
  Interventions: Behavioral: MBCT for Migraine
- Wait List/Treatment as Usual (No Intervention): Patients will continue with standard care. Patients will be offered MBCT after the primary endpoint.

INTERVENTIONS:
Behavioral: MBCT for Migraine — 8 75-90 minute individual sessions of the manualized Mindfulness-based Cognitive Therapy plus a manual and homework
  Arms: MBCT for Migraine

SUMMARY:
This randomized clinical trial aims to examine the effect of a standardized 8-week course of Mindfulness Based Cognitive Therapy for Migraine on migraine-related disability in people with migraine.

ELIGIBILITY:
Inclusion Criteria:

* ICHD-3 beta headache diagnosis of migraine,
* self-reported and diary-confirmed 4-20 headache days per month
* aged 18-65
* ability to read English
* capacity to consent.

Exclusion Criteria:

* no ICHD-3 beta headache diagnosis of migraine
* fewer than 4 or greater than 20 headache days per month
* under 18 or over 65
* inability to read English
* lacking the capacity to consent
* utilization of new preventative pain treatments within four weeks of the baseline assessment, or a plan to utilize new preventive pain medications during the duration of the study
* severe psychiatric illness that would interfere with participation in the treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Seng, Ph.D., Principal Investigator — Yeshiva University/Albert Einstein College of Medicine
Locations (1):
- Yeshiva University, The Bronx, New York, United States

REFERENCES:
- [Derived] Best RD, Ozmeral A, Grinberg AS, Smitherman TA, Seng EK. Pain acceptance as a change mechanism for mindfulness-based cognitive therapy for migraine. J Behav Med. 2024 Jun;47(3):471-482. doi: 10.1007/s10865-024-00475-5. Epub 2024 Feb 26. PMID 38407727
- [Derived] Seng EK, Conway AB, Grinberg AS, Patel ZS, Marzouk M, Rosenberg L, Metts C, Day MA, Minen MT, Buse DC, Lipton RB. Response to Mindfulness-Based Cognitive Therapy Differs Between Chronic and Episodic Migraine. Neurol Clin Pract. 2021 Jun;11(3):194-205. doi: 10.1212/CPJ.0000000000000984. PMID 34484887

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Started | 31 | 29
Completed | 29 | 26
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (10.6) | 44.2 (11.5) | 40.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 26 | 23 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60
Headache Disability Inventory (HDI) [Mean (Standard Deviation); unit: units on a scale] — The HDI is a scale that ranges from 0-100, with higher scores indicating higher levels of headache disability.
  units on a scale | 52.5 (21.2) | 50.2 (16.2) | 51.4 (19.0)
Migraine Disability Assessment (MIDAS) Score >=21 [Count of Participants; unit: Participants] — The MIDAS is a scale that assesses the number of days in the past three months participants experienced partially or fully reduced functioning in a variety of contexts (work, school, social). MIDAS scores are totaled and interpreted in the following grades: 0-5 = Grade I (Little or no disability); 6-10 = Grade II (Mild disability); 11-20 = Grade III (Moderate disability); 21+ = Grade IV (Severe disability). Scores were dichotomized at "Not Severe" (Grades I, II, and III) and "Severe "(Grade IV).
  Participants
    MIDAS Severe (Score >=21) | 24 | 26 | 50
    MIDAS Not Severe (Score < 21) | 7 | 3 | 10
Headache Day Frequency (>=15 days/30 days) [Count of Participants; unit: Participants]
  >= 15 days/month | 16 | 15 | 31
  < 15 days/month | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Proportion of People With "Severe" Scores on the Migraine Disability Assessment
Description: The MIDAS is a 5-item, self-report instrument that assesses the number of days in the past three months participants experienced partially or fully reduced functioning in a variety of contexts (work, school, social). MIDAS scores are totaled and interpreted in the following grades: 0-5 = Grade I (Little or no disability); 6-10 = Grade II (Mild disability); 11-20 = Grade III (Moderate disability); 21+ = Grade IV (Severe disability). Scores were dichotomized at "Not Severe" (Grades I, II, and III) and "Severe "(Grade IV). The outcome was the proportion of participants who reported "Severe Disability."
Time Frame: Change from Month 1 to Month 4
Measure: Number; unit: percentage of participants
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
percentage of participants
  Month 1 | 77.4 | 89.7
  Month 4 | 58.1 | 75.9
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .027, Mixed Models Analysis — Significance threshold set a priori at .025 to adjust for two co-primary outcomes; The key test was the Treatment (MBCT-M vs. WL.TAU) X Time (Month 1 vs 4) interaction with both Treatment and Time in the model; Slope = 1.6, 95% CI 2-sided [-0.7 to 3.9] — A positive slope indicates greater reduction in the proportino of people with Severe MIDAS scores (Score >=21) in the MBCT-M group vs. the WL/TAU group

2. Primary Outcome: Headache-Related Disability Index
Description: 25-item, self-report questionnaire of the emotional and functional impact of headache on daily activities. Total scores range from 0-100, with higher scores indicating higher levels of disability.
Time Frame: Change from Month 1 to Month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
score on a scale
  Month 1 | 52.5 (21.2) | 50.2 (16.2)
  Month 4 | 38.2 (16.6) | 50.4 (14.3)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p < .004, Mixed Models Analysis — Significance threshold set a priori at .025 to account for two co-primary outcomes; [statistical method as in outcome 1, analysis 1]; Slope = 14.1, 95% CI 2-sided [0.8 to 21.8] — Positive slope indicated larger reductions in HDI in the MBCT-M group compared to the WL/TAU group

3. Secondary Outcome: Headache Days (Over Course of 1 Month)
Description: Number of headache days/month for the month prior to treatment, and the month after treatment
Time Frame: Change from Month 1 to Month 4
Measure: Mean (Standard Deviation); unit: Days/30 days
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
Days/30 days
  Month 1 | 16.5 (6.0) | 15.5 (5.9)
  Month 4 | 14.8 (4.8) | 14.2 (4.8)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .773, Mixed Models Analysis — Threshold for statistical significance set a priori at .05; Key test was the Treatment (MBCT-M vs. WL/TAU) X Time (Month 1 vs. 4) interaction with Treatment and Time in the model; Slope = -.05, 95% CI 2-sided [-3.7 to 2.8] — A positive slope indicates greater reduction in headache days in the MBCT-M group vs. the WL/TAU group

4. Secondary Outcome: Average Headache Severity for Headache Days Recorded Over 30 Days
Description: Headache Severity was recorded for every headache day on a scale of 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe. Average headache severity was averaged across all headache days for each month.
Time Frame: Change from Month 1 to Month 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
units on a scale
  Month 1 | 1.7 (0.3) | 1.8 (0.3)
  Month 4 | 1.6 (0.3) | 1.7 (0.3)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .888, Mixed Models Analysis — Threshold for significance set a priori at .05; [statistical method as in outcome 1, analysis 1]; Slope = 0.01, 95% CI 2-sided [-0.14 to 0.16] — A positive slope indicates a greater reduction in headache attack pain intensity in the MBCT-M group vs. WL/TAU

5. Secondary Outcome: The Pain Catastrophizing Scale
Description: 13-item self-report measure that conveys a participant's level of pain-related, catastrophic thinking during painful experiences. Total scores range from 0-52, with higher scores indicating higher levels of catastrophizing.
Time Frame: Change from Month 1 to Month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
score on a scale
  Month 1 | 22.6 (8.7) | 22.0 (7.8)
  Month 4 | 15.6 (8.8) | 22.6 (10.4)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .035, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope = 7.45, 95% CI 2-sided [2.48 to 12.42] — A positive slope indicates a greater reduction in Pain Catastrophizing Scale in the MBCT-M group vs. WL/TAU

6. Secondary Outcome: Chronic Pain Acceptance Questionnaire
Description: 20-item, self-report measure of pain-related acceptance. Total scores range from 0-156 with higher scores indicating higher pain acceptance.
Time Frame: Change from Month 1 to Month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
score on a scale
  Month 1 | 60.7 (20.2) | 60.3 (14.0)
  Month 4 | 68.0 (9.2) | 64.7 (7.8)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .572, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope = -3.05, 95% CI 2-sided [-10.83 to 4.74] — A negative slope indicates a greater improvement in Chronic Pain Acceptance in the MBCT-M group vs. WL/TAU

7. Secondary Outcome: Five Facet Mindfulness Questionnaire
Description: 39-item self-report instrument assessing mindfulness. Total scores range from 39-195, with higher scores indicating higher levels of mindfulness.
Time Frame: Change from Month 1 to Month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
score on a scale
  Month 1 | 128.5 (17.6) | 132.9 (18.3)
  Month 4 | 116.0 (8.6) | 117.7 (10.9)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .609, Mixed Models Analysis — Threshold for significance set a priori at .05; [statistical method as in outcome 1, analysis 1]; Slope = -2.65, 95% CI 2-sided [-11.76 to 6.46] — A negative slope indicates a smaller decrease in the Five Factor Mindfulness Questionnaire in the MBCT-M group vs. WL/TAU

8. Secondary Outcome: Headache Specific Locus of Control
Description: 33-item measure designed to assess the extent to which individuals with recurrent headaches expect that the occurrence, worsening, and improvement of their headaches are influenced primarily by their own behavior, by chance or fate, or by the actions of medical professionals. Total scores range from 33-165, with higher scores indicating more external (vs. internal) locus of control.
Time Frame: Change from Month 1 to Month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
score on a scale
  Month 1 | 86.0 (10.5) | 87.5 (14.3)
  Month 4 | 80.3 (11.8) | 89.8 (17.1)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .022, Mixed Models Analysis — Threshold for significance set a priori at .05; [statistical method as in outcome 1, analysis 1]; Slope = 8.45, 95% CI 2-sided [2.99 to 13.91] — A positive slope indicates a greater reduction in Headache Specific Locus of Control Scale score in the MBCT-M group vs. WL/TAU

9. Secondary Outcome: Headache Management Self-efficacy Scale
Description: 25-item self-report scale designed to capture the confidence a patient believes they have in their own abilities to prevent headache episodes and manage their pain. Total scores range from 25-175, with higher scores indicating higher levels of self-efficacy
Time Frame: Change from Month 1 to Month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
score on a scale
  Month 1 | 108.1 (11.9) | 111.8 (13.5)
  Month 4 | 113.8 (12.6) | 115.4 (11.1)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .124, Mixed Models Analysis — Threshold for significance set a priori at .05; [statistical method as in outcome 1, analysis 1]; Slope = -2.01, 95% CI 2-sided [-7.56 to 3.53] — A negative slope indicates a greater improvement in Headache Management Self-Efficacy Scale score in the MBCT-M group vs. WL/TAU

10. Secondary Outcome: NIH PROMIS Depression Short Form
Description: 8-item self-report measure that assesses emotional distress in the past week focusing on negative mood and negative self-views. Scores are normed using T-scores (M = 50, SD = 10) with higher scores indicating higher levels of depressive symptoms.
Time Frame: Change from Month 1 to Month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
score on a scale
  Month 1 | 54.0 (60.2) | 53.1 (7.4)
  Month 4 | 52.2 (6.8) | 55.9 (6.5)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .017, Mixed Models Analysis — Threshold for significance set a priori at .05; [statistical method as in outcome 1, analysis 1]; Slope = 3.48, 95% CI 2-sided [0.63 to 6.33] — A positive slope indicates a greater reduction in PROMIS-Depression score in the MBCT-M group vs. WL/TAU

11. Secondary Outcome: NIH PROMIS Anxiety Short Form
Description: 8-item self-report measure that assesses emotional distress in the past week focusing on fear, worry and hyper-arousal. Scores were normed using T-scores (M = 50, SD = 10) with higher scores indicating higher levels of anxious symptoms.
Time Frame: Change from Month 1 to Month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
score on a scale
  Month 1 | 56.7 (8.2) | 56.2 (6.2)
  Month 4 | 55.7 (8.1) | 59.2 (7.7)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .259, Mixed Models Analysis — Threshold for significance set a priori at .05; [statistical method as in outcome 1, analysis 1]; Slope = 2.82, 95% CI 2-sided [-0.03 to 5.68] — A positive slope indicates a greater reduction in PROMIS-Anxiety score in the MBCT-M group vs. WL/TAU

12. Secondary Outcome: Average Monthly Migraine Disability Index
Description: A daily 4-item measure of migraine related disability. Scores range from 0-10, with higher scores indicating higher levels of disability. Scores are averaged across all headache days recorded each month.
Time Frame: Change from Month 1 through Month 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
Number analyzed (Participants) | 31 | 29
score on a scale
  Month 1 | 2.8 (1.6) | 3.4 (2.0)
  Month 4 | 1.7 (2.7) | 4.4 (1.3)
Statistical Analysis 1: Comparison: MBCT for Migraine vs Wait List/Treatment as Usual; Test type: Superiority; p = .007, Mixed Models Analysis; The key test was the Treatment (MBCT-M vs. WL/TAU) X Time (Month 1 vs. 4) interaction with both Treatment and Time in the model; Slope = -1.0, 95% CI 2-sided [-1.6 to -0.3] — A negative slope indicated a larger decrease in MIDI scores in the MBCT-M group vs. WL/TAU

ADVERSE EVENTS:
Time Frame: 4 months
Description: Adverse events were tracked on a monthly basis by research staff in both groups. Participants in the MBCT-M group were also tracked weekly by the study therapist during the two-month treatment period (Month 2 and Month 3).
Arm/Group | MBCT for Migraine | Wait List/Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 2/31 | 0/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBCT for Migraine (N=31) | Wait List/Treatment as Usual (N=29)
Flooding (Psychiatric disorders) | 1 (1) | 0 (0) — A vivid recollection of a traumatic event
Increase in headache frequency and intensity (Nervous system disorders) | 1 (1) | 0 (0) — Sudden and severe increase in headache frequency and intensity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT02443519/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT02443519/ICF_001.pdf